CLINICAL TRIAL: NCT05995353
Title: A Phase 3, Multi-Center Study to Evaluate the Pharmacokinetics, Efficacy, and Safety of Risankizumab With Open-Label Induction, Randomized Double-Blind Maintenance, and Long-Term Extension Periods in Pediatric Subjects (2 to < 18 Years of Age) With Moderately to Severely Active Crohn's Disease
Brief Title: A Study to Assess Adverse Events, Change in Disease Activity, and How Intravenous and Subcutaneous Risankizumab Moves Through the Body of Pediatric Participants With Moderately to Severely Active Crohn's Disease
Acronym: RISE
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: M16-194; 2022-502050-14-00 (Other: EU CT)
Record Dates: First submitted 2023-08-10; First posted 2023-08-16 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Crohn's Disease
Keywords: Crohn's Disease; Risankizumab; Skyrizi; Pediatrics
MeSH Terms: conditions — Crohn Disease | interventions — risankizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (15):
- PK Cohort 1: SS1 (Experimental): Cohort 1 (including Sub-cohort 1A) will consist of 2 age groups (6 to < 12 years and 12 to < 18 years). SS1 is a 12-week induction period where participants will receive a weight-based dose of risankizumab. All participants who complete SS1 are eligible to enter SS2.
  Interventions: Drug: Risankizumab
- PK Cohort 1: SS2 Dose A (Experimental): Cohort 1 (including Sub-cohort 1A) will consist of 2 age groups (6 to < 12 years and 12 to < 18 years). Participants who complete SS1 will be randomized into a 52-week maintenance phase (SS2) to receive double-blind risankizumab Dose A. Participants who complete SS2 will have the opportunity to enter the open-label long-term-extension SS3.
  Interventions: Drug: Risankizumab
- PK Cohort 1: SS2 Dose B (Experimental): Cohort 1 (including Sub-cohort 1A) will consist of 2 age groups (6 to < 12 years and 12 to < 18 years). Participants who complete SS1 will be randomized into a 52-week maintenance phase (SS2) to receive double-blind risankizumab Dose B. Participants who complete SS2 will have the opportunity to enter the open-label long-term-extension SS3.
  Interventions: Drug: Risankizumab
- PK Cohort 1: SS3 Dose A (Experimental): Cohort 1 (including Sub-cohort 1A) will consist of 2 age groups (6 to < 12 years and 12 to < 18 years). SS3 is a 208-week extension period where participants receive risankizumab based on their response in SS2.
  Interventions: Drug: Risankizumab
- PK Cohort 1: SS3 Dose B (Experimental): Cohort 1 (including Sub-cohort 1A) will consist of 2 age groups (6 to < 12 years and 12 to < 18 years). SS3 is a 208-week extension period where participants receive risankizumab based on their response in SS2.
  Interventions: Drug: Risankizumab
- PK Cohort 2: SS1 (Experimental): Cohort 2 will enroll participants aged 2 to less than 6 years. SS1 is a 12-week induction period where participants will receive a weight-based dose of risankizumab. All subjects who complete SS1 are eligible to enter SS2.
  Interventions: Drug: Risankizumab
- PK Cohort 2: SS2 Dose A (Experimental): Cohort 2 will enroll participants aged 2 to less than 6 years. Participants who complete SS1 will be randomized into a 52-week maintenance phase (SS2) to receive double-blind risankizumab Dose A. Participants who complete SS2 will have the opportunity to enter the open-label long-term-extension SS3.
  Interventions: Drug: Risankizumab
- PK Cohort 2: SS2 Dose B (Experimental): Cohort 2 will enroll participants aged 2 to less than 6 years. Participants who complete SS1 will be randomized into a 52-week maintenance phase (SS2) to receive double-blind risankizumab Dose B. Participants who complete SS2 will have the opportunity to enter the open-label long-term-extension SS3.
  Interventions: Drug: Risankizumab
- PK Cohort 2: SS3 Dose A (Experimental): Cohort 2 will enroll participants aged 2 to less than 6 years. SS3 is a 208-week extension period where participants receive risankizumab based on their response in SS2.
  Interventions: Drug: Risankizumab
- PK Cohort 2: SS3 Dose B (Experimental): Cohort 2 will enroll participants aged 2 to less than 6 years. SS3 is a 208-week extension period where participants receive risankizumab based on their response in SS2.
  Interventions: Drug: Risankizumab
- Expansion Cohort 3: SS1 (Experimental): Cohort 3 will enroll participants aged 2 to less than 18 years. SS1 is a 12-week induction period where participants will receive a weight-based dose of risankizumab. All subjects who complete SS1 are eligible to enter SS2.
  Interventions: Drug: Risankizumab
- Expansion Cohort 3: SS2 Dose A (Experimental): Cohort 3 will enroll participants aged 2 to less than 18 years. Participants who complete SS1 will be randomized into a 52-week maintenance phase (SS2) to receive either double-blind risankizumab Dose A. Participants who complete SS2 will have the opportunity to enter the open-label long-term-extension SS3.
  Interventions: Drug: Risankizumab
- Expansion Cohort 3: SS2 Dose B (Experimental): Cohort 3 will enroll participants aged 2 to less than 18 years. Participants who complete SS1 will be randomized into a 52-week maintenance phase (SS2) to receive either double-blind risankizumab Dose B. Participants who complete SS2 will have the opportunity to enter the open-label long-term-extension SS3.
  Interventions: Drug: Risankizumab
- Expansion Cohort 3: SS3 Dose A (Experimental): Cohort 3 will enroll participants aged 2 to less than 18 years. SS3 is a 208-week extension period where participants receive risankizumab based on their response in SS2.
  Interventions: Drug: Risankizumab
- Expansion Cohort 3: SS3 Dose B (Experimental): Cohort 3 will enroll participants aged 2 to less than 18 years. SS3 is a 208-week extension period where participants receive risankizumab based on their response in SS2.
  Interventions: Drug: Risankizumab

INTERVENTIONS:
Drug: Risankizumab — Intravenous (IV) Infusion
  Other Names: ABBV-066; SKYRIZI
  Arms: Expansion Cohort 3: SS1; PK Cohort 1: SS1; PK Cohort 2: SS1
Drug: Risankizumab — Subcutaneous (SC) Injection
  Other Names: ABBV-066; SKYRIZI
  Arms: Expansion Cohort 3: SS2 Dose A; Expansion Cohort 3: SS2 Dose B; Expansion Cohort 3: SS3 Dose A; Expansion Cohort 3: SS3 Dose B; PK Cohort 1: SS2 Dose A; PK Cohort 1: SS2 Dose B; PK Cohort 1: SS3 Dose A; PK Cohort 1: SS3 Dose B; PK Cohort 2: SS2 Dose A; PK Cohort 2: SS2 Dose B; PK Cohort 2: SS3 Dose A; PK Cohort 2: SS3 Dose B

SUMMARY:
Crohn's Disease (CD) is a gastrointestinal disease that can cause chronic diarrhea with or without gross bleeding, abdominal pain, weight loss, and fever. This study will assess the pharmacokinetics, efficacy, and safety of risankizumab in pediatric participants with moderately to severely active CD aged 2 to < 18 years old who have had intolerance or inadequate response to other therapies.

Risankizumab is an approved drug for adults with plaque psoriasis, psoriatic arthritis, and CD and is being developed for the treatment of CD in pediatrics. This study is comprised of 3 cohorts that may participate in 3 substudies (SS). Cohort 1(including Sub-cohort 1A) will enroll participants with ages from 6 to less than 18 years. Cohort 2 will enroll participants with ages from 2 to less than 6 years. Cohort 3 will enroll participants with ages from 2 to less than 18 years. SS1 is an open-label induction period where participants will receive a weight-based induction regimen of risankizumab. SS2 is a double-blind maintenance period where participants will be randomized to receive 1 of 2 doses of weight-based induction regimen of risankizumab. SS3 is an open-label extension period where participants will receive risankizumab based off of their response in SS2. Approximately 118 pediatric participants with CD will be enrolled at around 100 sites worldwide.

Participants in SS1 will receive risankizumab intravenously during the 12-week induction period. Participants in SS2 will receive risankizumab subcutaneously during the 52-week randomized maintenance period. Participants in SS3 will receive risankizumab subcutaneously during the 208-week open label period. Participants will be followed-up for approximately 140 days.

There may be higher treatment burden for participants in this trial compared to their standard of care. Participants will attend regular visits during the study at a hospital or clinic. The effect of the treatment will be checked by medical assessments, blood tests, checking for side effects and completing questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric individuals, 2 to < 18 years old
* Must have moderately to severely active CD, as defined by the PCDAI score > 30 assessed at Baseline
* Must have endoscopic evidence of mucosal inflammation as documented by the SES-CD of ≥ 6 for ileocolonic or colonic disease (or SES-CD of ≥ 4 for isolated ileal disease)
* Demonstrated intolerance or inadequate response to one or more of the following categories of drugs: aminosalicylates (This drug class is not sufficient for eligibility for subjects in France, Italy, Netherlands, Spain, and Sweden), oral locally acting corticosteroids, systemic steroids (prednisone or equivalent), IMMs, and/or biologic therapies

Exclusion Criteria:

* History of hereditary fructose intolerance (a rare genetic condition) or an allergic reaction or significant sensitivity to constituents of the study drug (and its excipients) and/or other products in the same class
* Any of the following medical disorders:

  1. Current diagnosis of ulcerative colitis, indeterminate colitis, or monogenic IBD.
  2. A diagnosis of CD prior to 2 years of age.
  3. A diagnosis or suspected diagnosis of a primary immunodeficiency.
  4. Currently known complications of CD such as:

     * Active abscess (abdominal or perianal);
     * Symptomatic bowel strictures;
     * > 2 missing segments of the following 5 segments: terminal ileum, right colon, transverse colon, sigmoid and left colon, and rectum;
     * Fulminant colitis;
     * Toxic megacolon;
     * Or any other manifestation that might require surgery while enrolled in the study.
  5. Ostomy or ileoanal pouch.
  6. Diagnosis of short gut or short bowel syndrome.
  7. Surgical bowel resection within the past 3 months prior to Baseline (excluding gastrointestinal surgeries which are not bowel resections such as appendectomy or ostomy closure), or a history of >3 bowel resections.

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 118 (Estimated)
Dates: Start 2023-12-11 (Actual); Primary Completion 2029-04 (Estimated); Study Completion 2029-04 (Estimated)

PRIMARY OUTCOMES:
Cohort 3 (Substudy 2): Percentage of Participants Achieving Pediatric Crohn's Disease Activity Index (PCDAI) Clinical Remission | At 64 weeks
  PCDAI is an index used to measure disease activity of pediatric patients with Crohn's disease assessing abdominal pain, stool frequency, patient functioning, hematocrit, erythrocyte sedimentation rate, albumin, weight, height, abdomen, perirectal disease, and extraintestinal manifestations. It ranges from 0 to 100; higher scores indicate more active disease. Clinical remission was defined as PCDAI ≤ 10.
Cohort 3 (Substudy 2): Percentage of Participants Achieving Endoscopic Response per Simple Endoscopic Score for Crohn's Disease (SES-CD) | At 64 weeks
  The SES-CD assesses endoscopic disease severity by evidence of active intestinal mucosal inflammation. Endoscopic response is defined as a decrease in SES-CD > 50% from Baseline (or for participants with isolated ileal disease and a Baseline SES-CD of 4, at least a 2-point reduction from Baseline).
Cohorts 1 & 2: Maximum Observed Serum Concentration (Cmax) of Risankizumab | Up to approximately Week 64
  Cmax of risankizumab
Cohorts 1 & 2: Time to Cmax (Tmax) of Risankizumab | Up to approximately 64 weeks
  Tmax of risankizumab
Cohorts 1 & 2: Area Under the Serum Concentration-Time Curve Over the Dosing Interval (AUCtau) of Risankizumab | Up to approximately 64 weeks
  AUCtau of risankizumab

SECONDARY OUTCOMES:
Cohort 3 (Substudy 1): Percentage of Participants Achieving PCDAI Clinical Remission | At 12 weeks
  PCDAI is an index used to measure disease activity of pediatric patients with Crohn's disease assessing abdominal pain, stool frequency, patient functioning, hematocrit, erythrocyte sedimentation rate, albumin, weight, height, abdomen, perirectal disease, and extraintestinal manifestations. It ranges from 0 to 100; higher scores indicate more active disease. Clinical remission was defined as PCDAI ≤ 10.
Cohort 3 (Substudy 1): Percentage of Participants Achieving Endoscopic Response per SES-CD | At 12 weeks
  The SES-CD assesses endoscopic disease severity by evidence of active intestinal mucosal inflammation. Endoscopic response is defined as a decrease in SES-CD > 50% from Baseline (or for participants with isolated ileal disease and a Baseline SES-CD of 4, at least a 2-point reduction from Baseline).
Cohort 3 (Substudy 1): Percentage of Participants Achieving Endoscopic Remission per SES-CD | At 12 weeks
  The SES-CD assesses endoscopic disease severity by evidence of active intestinal mucosal inflammation. Endoscopic remission is defined as SES-CD ≤ 4 with at least a 2-point reduction from Baseline and no sub-score > 1, as scored by a central reader.
Cohort 3 (Substudy 2): Percentage of Participants Achieving Endoscopic Remission per SES-CD | At 64 weeks
  The SES-CD assesses endoscopic disease severity by evidence of active intestinal mucosal inflammation. Endoscopic remission is defined as SES-CD ≤ 4 with at least a 2-point reduction from Baseline and no sub-score > 1, as scored by a central reader.
Cohort 3 (Substudy 2): Percentage of Participants Achieving Corticosteroid-Free Clinical Remission per PCDAI | At 64 weeks
  PCDAI is an index used to measure disease activity of pediatric patients with Crohn's disease assessing abdominal pain, stool frequency, patient functioning, hematocrit, erythrocyte sedimentation rate, albumin, weight, height, abdomen, perirectal disease, and extraintestinal manifestations. It ranges from 0 to 100; higher scores indicate more active disease. PCDAI corticosteroid-free remission was defined as discontinued corticosteroid use at least 90 consecutive days prior to the respective visit, with a PCDAI ≤ 10 at that visit.
Cohorts 1 & 2 (Substudy 2): Percentage of Participants Achieving PCDAI Clinical Remission | At 64 weeks
  PCDAI is an index used to measure disease activity of pediatric patients with Crohn's disease assessing abdominal pain, stool frequency, patient functioning, hematocrit, erythrocyte sedimentation rate, albumin, weight, height, abdomen, perirectal disease, and extraintestinal manifestations. It ranges from 0 to 100; higher scores indicate more active disease. Clinical remission was defined as PCDAI ≤ 10.
Cohorts 1 & 2 (Substudy 2): Percentage of Participants Achieving Endoscopic Response per SES-CD | At 64 weeks
  The SES-CD assesses endoscopic disease severity by evidence of active intestinal mucosal inflammation. Endoscopic response is defined as a decrease in SES-CD > 50% from Baseline (or for participants with isolated ileal disease and a Baseline SES-CD of 4, at least a 2-point reduction from Baseline).
Cohorts 1 & 2 (Substudy 1): Percentage of Participants Achieving PCDAI Clinical Remission | At 12 weeks
  PCDAI is an index used to measure disease activity of pediatric patients with Crohn's disease assessing abdominal pain, stool frequency, patient functioning, hematocrit, erythrocyte sedimentation rate, albumin, weight, height, abdomen, perirectal disease, and extraintestinal manifestations. It ranges from 0 to 100; higher scores indicate more active disease. Clinical remission was defined as PCDAI ≤ 10.
Cohorts 1 & 2 (Substudy 1): Percentage of Participants Achieving Endoscopic Response per SES-CD | At 12 weeks
  The SES-CD assesses endoscopic disease severity by evidence of active intestinal mucosal inflammation. Endoscopic response is defined as a decrease in SES-CD > 50% from Baseline (or for participants with isolated ileal disease and a Baseline SES-CD of 4, at least a 2-point reduction from Baseline).
Cohorts 1 & 2 (Substudy 1): Percentage of Participants Achieving Endoscopic Remission per SES-CD | At 12 weeks
  The SES-CD assesses endoscopic disease severity by evidence of active intestinal mucosal inflammation. Endoscopic remission is defined as SES-CD ≤ 4 with at least a 2-point reduction from Baseline and no sub-score > 1, as scored by a central reader.
Cohorts 1 & 2 (Substudy 2): Percentage of Participants Achieving Endoscopic Remission per SES-CD | At 64 weeks
  The SES-CD assesses endoscopic disease severity by evidence of active intestinal mucosal inflammation. Endoscopic remission is defined as SES-CD ≤ 4 with at least a 2-point reduction from Baseline and no sub-score > 1, as scored by a central reader.
Cohorts 1 & 2 (Substudy 2): Percentage of Participants Achieving Corticosteroid-Free Clinical Remission per PCDAI | At 64 weeks
  PCDAI is an index used to measure disease activity of pediatric patients with Crohn's disease assessing abdominal pain, stool frequency, patient functioning, hematocrit, erythrocyte sedimentation rate, albumin, weight, height, abdomen, perirectal disease, and extraintestinal manifestations. It ranges from 0 to 100; higher scores indicate more active disease. PCDAI corticosteroid-free remission was defined as discontinued corticosteroid use at least 90 consecutive days prior to the respective visit, with a PCDAI ≤ 10 at that visit.

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (85):
- United States (11):
  - Phoenix Children's Hospital /ID# 255766, Phoenix, Arizona
  - Arkansas Children's Hospital /ID# 255762, Little Rock, Arkansas
  - UCSF Benioff Children's Hospital - Oakland /ID# 258327, Oakland, California
  - Children's Hospital Colorado - Aurora /ID# 255764, Aurora, Colorado
  - Arnold Palmer Hospital for Children Center Digestive Health & Nutrition - Orland /ID# 255437, Orlando, Florida
  - Indiana University Health Riley Hospital for Children /ID# 256454, Indianapolis, Indiana
  - Massachusetts General Hospital /ID# 255767, Boston, Massachusetts
  - MNGI Digestive Health, P. A. /ID# 255366, Minneapolis, Minnesota
  - Goryeb Childrens Hospital /ID# 256452, Morristown, New Jersey
  - Icahn School of Medicine at Mount Sinai /ID# 254880, New York, New York
  - Cleveland Clinic - Cleveland /ID# 256453, Cleveland, Ohio
- Belgium (6):
  - Uza /Id# 255114, Edegem, Antwerpen
  - Cliniques Universitaires UCL Saint-Luc /ID# 255108, Brussels, Brussels Capital
  - Universitair Ziekenhuis Brussel /ID# 255109, Jette, Brussels Capital
  - Groupe Sante CHC - Clinique du MontLegia /ID# 255620, Liège, Liege
  - Universitair Ziekenhuis Leuven /ID# 255098, Leuven, Vlaams-Brabant
  - Hospital Universite Enfants Reine Fabiola /ID# 255112, Brussels
- Bulgaria (3):
  - UMHAT Sveti Georgi /ID# 255386, Plovdiv
  - Specialized Hospital For Active Treatment Of Children Diseases Prof. Ivan Mitev /ID# 255384, Sofia
  - UMHAT Multiprofile Hospital for Active Treatment Sveta Marina /ID# 256358, Varna
- Canada (4):
  - Alberta Children's Hospital /ID# 255357, Calgary, Alberta
  - Edmonton Clinic Health Academy /ID# 255361, Edmonton, Alberta
  - BC Children's Hospital /ID# 255359, Vancouver, British Columbia
  - London Health Sciences Centre - Victoria Hospital & Children's Hospital /ID# 258598, London, Ontario
- China (10):
  - Beijing Children's Hospital /ID# 256081, Beijing, Beijing Municipality
  - Peking University Third Hospital /ID# 255876, Beijing, Beijing Municipality
  - Guangzhou Medical University Affiliated Women and Children's Medical Center /ID# 255428, Guangzhou, Guangdong
  - The Sixth Affiliated Hospital of Sun Yat-sen University /ID# 270589, Guangzhou, Guangdong
  - Henan Children's Hospital Zhengzhou Children's Hospital /ID# 255562, Zhengzhou, Henan
  - Hunan Children's Hospital /ID# 255610, Changsha, Hunan
  - Jiangxi Provincial Children's Hospital /ID# 255564, Nanchang, Jiangxi
  - Shengjing Hospital of China Medical University /ID# 255563, Shenyang, Liaoning
  - Children's Hospital of Shanghai /ID# 255531, Shanghai, Shanghai Municipality
  - Ruijin Hospital, Shanghai Jiaotong University School of Medicine /ID# 255688, Shanghai, Shanghai Municipality
- Czechia (2):
  - Vseobecna Fakultni Nemocnice v Praze /ID# 256096, Prague, Praha 17
  - Fakultní nemocnice v Motole /ID# 256547, Prague, Praha 5
- France (5):
  - CHRU Tours - Hopital Gatien de Clocheville /ID# 255052, Tours, Centre-Val de Loire
  - CHU Bordeaux - Hopital Pellegrin /ID# 257060, Bordeaux, Nouvelle-Aquitaine
  - Hospices Civils de Lyon - Hôpital Femme Mère Enfant /ID# 255443, Bron, Rhone
  - AP-HP - Hopital Necker /ID# 255608, Paris
  - CHU Toulouse - Hopital Paule de Viguier /ID# 255609, Toulouse
- Germany (2):
  - Dr. von Haunerschen Kinderspital /ID# 255577, Munich, Bavaria
  - Universitaetsklinikum Muenster /ID# 256762, Münster, North Rhine-Westphalia
- Israel (2):
  - Schneider Children's Medical Center /ID# 254950, Petah Tikva, Central District
  - Shaare Zedek Medical Center /ID# 254951, Jerusalem, Jerusalem
- Italy (4):
  - IRCCS Istituto Giannina Gaslini /ID# 255262, Genoa, Genova
  - Azienda Ospedaliera Universitaria Federico II /ID# 255045, Naples, Napoli
  - Ospedale Pediatrico Bambino Gesù /ID# 255043, Rome, Roma
  - Azienda Ospedaliera Universitaria Gaetano Martino /ID# 255044, Messina
- Japan (10):
  - Aichi Children'S Health And Medical Center /ID# 272085, Ōbu, Aichi-ken
  - Tsujinaka Hospital - Kashiwanoha /ID# 268409, Kashiwa-shi, Chiba
  - Kurume University Hospital /ID# 268418, Kurume-shi, Fukuoka
  - Gunma University Hospital /ID# 270560, Maebashi, Gunma
  - Japanese Red Cross Kumamoto Hospital /ID# 268586, Kumamoto, Kumamoto
  - Osaka Women's and Children's Hospital /ID# 268419, Izumi-Shi, Osaka
  - Saitama Children's Medical Center /ID# 268410, Saitama-shi, Saitama
  - Institute of Science Tokyo Hospital /ID# 269175, Bunkyo-ku, Tokyo
  - Tokyo Metropolitan Children's Medical Center /ID# 268415, Fuchu-shi, Tokyo
  - National Center For Child Health And Development /ID# 268420, Setagaya City, Tokyo
- Amsterdam UMC, locatie AMC /ID# 254827, Amsterdam, North Holland, Netherlands
- Poland (2):
  - Gastromed Sp. z o.o /ID# 255939, Torun, Kuyavian-Pomeranian Voivodeship
  - Instytut Pomnik - Centrum Zdrowia Dziecka /ID# 255938, Warsaw, Masovian Voivodeship
- Puerto Rico (2):
  - Puerto Rico Health Institute /ID# 255071, Dorado
  - Clinical Research Puerto Rico /ID# 266479, San Juan
- South Korea (4):
  - Seoul National University Hospital /ID# 255318, Seoul, Seoul Teugbyeolsi
  - Yonsei University Health System Severance Hospital /ID# 256976, Seoul, Seoul Teugbyeolsi
  - Samsung Medical Center /ID# 255284, Seoul, Seoul Teugbyeolsi
  - Kyungpook National University Chilgok Hospital /ID# 255817, Daegu
- Spain (3):
  - Hospital Arquitecto Marcide - Complejo Hospitalario Universitario de Ferrol /ID# 255614, Ferrol, A Coruna
  - Hospital Infantil Universitario Nino Jesus /ID# 255012, Madrid
  - Hospital Regional Universitario de Malaga /ID# 257553, Málaga
- Sweden (3):
  - Karolinska University Hospital Solna /ID# 255240, Solna, Stockholm County
  - Sodersjukhuset /ID# 255239, Stockholm, Stockholm County
  - Sahlgrenska Universitetssjukhuset /ID# 255236, Gothenburg, Västra Götaland County
- Switzerland (2):
  - University Children's Hospital Zurich - Eleonorenstiftung /ID# 255337, Zurich, Canton of Zurich
  - Inselspital, Universitaetsspital Bern /ID# 255321, Bern
- Taiwan (2):
  - National Taiwan University Hospital /ID# 255679, Taipei City, Taipei
  - Changhua Christian Hospital /ID# 256082, Changhua City, Changhua County
- Turkey (Türkiye) (4):
  - Gazi University Medical Faculty /ID# 255086, Ankara
  - Sariyer Hamidiye Etfal Eğitim Ve Araştirma Hastanesi /ID# 257143, Istanbul
  - Marmara Universitesi Pendik Egitim ve Arastirma Hastanesi /ID# 261020, Istanbul
  - Kocaeli University Med Faculty /ID# 256922, Kocaeli
- United Kingdom (3):
  - Sheffield Children's Hospital NHS Foundation Trust /ID# 255758, Sheffield, England
  - Disc_Barts Health NHS Trust - The Royal London Hospital /ID# 255757, London, Greater London
  - Birmingham Women's and Children's NHS Foundation Trust /ID# 255759, Birmingham

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible clinical trial data sharing. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information.
Supporting Information: Study Protocol, SAP
Time Frame: For details on when studies are available for sharing visit https://vivli.org/ourmember/abbvie/
Access Criteria: To learn more about the process, or to submit a request, visit the following link https://www.abbvieclinicaltrials.com/hcp/data-sharing/
URL: https://vivli.org/ourmember/abbvie/

REFERENCES:
- See also: Related Info — https://www.abbvieclinicaltrials.com/study/?id=M16-194